CLINICAL TRIAL: NCT03907514
Title: Impact of the Use of Digital Technology in Adolescent-dentist Interaction: Randomized Clinical Trial
Brief Title: Improving Adolescent-dentist Interaction Through Digital Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Trícia Murielly Andrade de Souza Mayer, PhD student in Pediatric Dentistry, Principal Investigator, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 022019
Record Dates: First submitted 2019-01-31; First posted 2019-04-09 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Dental Anxiety
Keywords: Technology Assessment, Health; Dental anxiety; Adolescent; Clinical Trial

STUDY DESIGN:
Masking Description: Blindness will be possible to the psychologist, who will evaluates the patient's cooperation, and the statistician responsible for the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): The adolescents in this group will use the "FALE" application through a smartphone in the waiting room before the dental appointment. When starting to answer the application, the adolescent will report his/her level of dental anxiety through the question, "How do you feel about coming to see your dentist today?", and record his/her answer on a seven-point face scale. Then the participant will continue to answer the 12 other questions, and finally registers his/her anxiety level once more through the same question.
  Interventions: Behavioral: "FALE" Application
- Control Group (CG) (No Intervention): Similarly to IG, the adolescents in this group will use the "FALE" application through a smartphone, but only to record their level of anxiety by answering the question "How do you feel about coming to see your dentist today?" using a seven-point face scale. Instead of continuing to answer the other questions, the application will guide him to wait for the one-minute interval (expected time to answer the questionnaire) and, once more, ask the same question regarding his/her feeling about the experience with the dentist.

INTERVENTIONS:
Behavioral: "FALE" Application — "FALE" is a digital tool, in the form of an application for smartphones, which aims to demonstrate empathy and facilitate communication between the adolescent patient and the dentist. The application contains 14 questions regarding dental anxiety, feelings and patient coping preferences regarding dental care.
  Arms: Intervention Group (IG)

SUMMARY:
The aim of the present study is to assess the impact of a digital tool on the interaction between the dentist and the adolescent patient, concerning the level of dental anxiety and communication. To achieve this purpose, a Randomized Controlled Clinical Trial will be performed using a short version of e-SAID (Survey of Anxiety and Information for Dentists) in Portuguese (FALE). That is, the intervention to be tested is an application usage, which will contain a questionnaire with questions supposedly made by the dentist, about feelings regarding the dental appointment and preferences for coping with dental treatment. Thus, the use of this digital tool aims to facilitate communication, favoring the adolescent-dentist relationship, and establishing empathy.

DETAILED DESCRIPTION:
The target population consists of patients between 10 and 19 years old, attending the Adolescent Clinic in the Dental School of the Federal University of Pernambuco (UFPE), campus of Recife. The sample will consist of 184 adolescents, 92 in each group (intervention and control). Randomization will be stratified according to sex, age and presence or absence of dental anxiety. In the waiting room, before the dental appointment, the adolescents in the intervention group (IG) will use the FALE application to answer the questionnaire and assess the level of anxiety. Those in the control group (CG) will only record their level of anxiety. The undergraduates responsible for attending the IG participants will receive, prior to dental care, a report of the answers given by the adolescents through the application. During the dental consultation, a psychologist, who will be observing the care, will evaluate the adolescents behavior, considering cooperation. After the appointment, the adolescent will evaluate how much he/she felt benefited by the use of the app; how he evaluates the communication between him/her and the dentist; if he/she thinks that the app contributed with this communication; his/her satisfaction with dental treatment; and his/her satisfaction with the undergraduate attendance. The undergraduate will also evaluate his/her level of satisfaction with the application's use; how he/she evaluates the communication between him/her and the adolescent patient; how much the application has helped with this communication; and the degree of patient's cooperation during the dental consultation. Descriptive and inferential statistical analysis will be performed using appropriate tests through the Statistical Package for Social Sciences software version 21 and significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian adolescents literate in Portuguese
* Brazilian adolescents able to use smartphone

Exclusion Criteria:

* Adolescents with intellectual, sensory or physical disabilities
* Adolescents not capable to read and write/type

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Changes in adolescent patient's level of dental anxiety through the FALE application. | The outcome measure will be assessed before a single dental appointment in two stages: at the beginning and after four minutes, in the end of the "FALE" application use.
  Changes in patient's level of dental anxiety will be obtained through the question: "How do you feel about coming to see your dentist today?". This question is inserted in the FALE application and is answered through a seven-point face scale.

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Colares, Professor, Study Chair — University of Pernambuco; Trícia Mayer, PhD student, Principal Investigator — University of Pernambuco
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yee R, Jones LM, Hosey MT. What the child "SAID" to the dentist: A UK randomized controlled trial. Child Care Health Dev. 2017 Nov;43(6):926-932. doi: 10.1111/cch.12510. Epub 2017 Aug 30. PMID 28857237
- [Background] Jones L. Validation and randomized control trial of the e-SAID, a computerized paediatric dental patient request form, to intervene in dental anxiety. Child Care Health Dev. 2015 Jul;41(4):620-5. doi: 10.1111/cch.12200. Epub 2014 Oct 6. PMID 25287626
- [Background] Jones LM, Huggins TJ. The rationale and pilot study of a new paediatric dental patient request form to improve communication and outcomes of dental appointments. Child Care Health Dev. 2013 Nov;39(6):869-72. doi: 10.1111/j.1365-2214.2012.01416.x. Epub 2012 Jul 30. PMID 22846104